CLINICAL TRIAL: NCT01526148
Title: Comparative Safety, Tolerability, and Effectiveness of Lithium Versus Quetiapine in Patients Across the Spectrum of Bipolar Disorder
Brief Title: Gao Bipolar Spectrum Lithium/Quetiapine Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Ran out of funding
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Keming Gao, Director, Mood & Anxiety Clinic, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-11-01
Record Dates: First submitted 2012-01-25; First posted 2012-02-03 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium (Active Comparator)
  Interventions: Drug: Lithium
- Quetiapine (Active Comparator)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Lithium — Lithium will be initiated at 300 mg per day and titrated in 300 mg increments every 7days as tolerated with blood lithium levels > 0.6mEq/L.
  Other Names: Lithium Carbonate; Eskalith
  Arms: Lithium
Drug: Quetiapine — Quetiapine will be started at 50 mg per day at bedtime and titrated up to 300 mg as tolerated over 1 week.
  Other Names: Seroquel
  Arms: Quetiapine

SUMMARY:
This is a 4-month randomized open-label comparative safety, tolerability, and effectiveness trial of Lithium versus Quetiapine for subjects presenting in any phase of Bipolar who currently require a medication change for their illness. Stratified randomization will reduce bipolar type I , bipolar type II , or sub-threshold imbalance across cells. The enrollment goal is 60 subjects, over 24 months from initial regulatory approval. The primary outcome is the difference between lithium and quetiapine in the time to 'all cause' medication discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent before beginning any study-specific procedures
* Male and female patients at least 18 years of age
* Meets Diagnostic and Statistical Manual -IV criteria for BPI, BP II, or National Comorbidity Survey-R criteria for sub-threshold BP with or without symptoms, in need of medication adjustment(s)
* Willing to be randomized to either Lithium or Quetiapine
* If a sexually active female of childbearing potential, be using a reliable method of contraception, such as oral contraceptive or long-term injectable or implantable hormonal contraceptive, double-barrier methods (e.g. condom and diaphragm, condom and foam, condom and sponge), intrauterine devices, and tubal ligation
* Women with reproductive potential must have a negative urine pregnancy test

Exclusion Criteria:

* Unwilling to comply with study requirements
* Patients who have had severe adverse reaction to Lithium or Quetiapine
* Patients who require inpatient care
* Drug/alcohol dependence requiring immediate acute detoxification
* Pregnancy as determined by serum pregnancy test or breastfeeding
* History of nonresponse to Lithium at doses >900 mg ≥8 wks or to Quetiapine at doses of at least 300 mg/d ≥ 8 week for depression and at least 400-600 mg/d ≥ 4 wks for mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center - Mood Disorders Program, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lithium | Quetiapine
Started | 18 | 24
Completed | 4 | 11
Not Completed | 14 | 13
Not completed — Adverse Event | 6 | 5
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Unstable Medical Condition | 1 | 0
Not completed — Unable to discontinue concomitant med | 1 | 0
Not completed — Moved out of state | 1 | 0
Not completed — Incarcerated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium | Quetiapine | Total
Number analyzed (Participants) | 18 | 24 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.26 (16.66) | 35.58 (12.64) | 38.98 (14.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 7 | 14 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 15 | 22
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Diagnosis [Number; unit: participants]
  Bipolar I Disorder | 10 | 15 | 25
  Bipolar II Disorder | 9 | 7 | 16
  Bipolar NOS | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Study Discontinuation
Description: The time, as measured in number of days, for discontinuation due to all causes will be measured and used as the primary outcome measure
Time Frame: Week 16
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Lithium | Quetiapine
Number analyzed (Participants) | 18 | 24
days | 41 [23 to 83] | 77 [38 to 200]

2. Secondary Outcome: Lithium vs. Quetiapine Effects on General Cardiovascular Disease Risk as Measured by Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Description: Change in homeostatic model assessment for insulin resistance (HOMA-IR) from screening to end of study. Insulin resistance is a condition in which cells fail to respond to the normal actions of the hormone in the body. The HOMA-IR is calculated using a subject's fasting plasma insulin and glucose levels. The higher the score, the higher the level of insulin resistance.
Time Frame: Screening and Week 16
Measure: Mean (Standard Deviation); unit: IR Score
Arm/Group | Lithium | Quetiapine
Number analyzed (Participants) | 18 | 24
IR Score | -5.5 (15.9) | 0.2 (1.6)

ADVERSE EVENTS:
Arm/Group | Lithium | Quetiapine
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/24
Other Adverse Events (participants affected / at risk) | 16/18 | 21/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=18) | Quetiapine (N=24)
Excessive sleepiness / daytime somnolence (General disorders) | 7 (7) | 12 (12)
Stomach Upset (Gastrointestinal disorders) | 5 (5) | 0 (0)
Increased thirst (General disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Insomnia (General disorders) | 3 (3) | 0 (0)
Increased urination (Renal and urinary disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 3 (3)
Headache (General disorders) | 2 (2) | 2 (2)
Muscle Stiffness (General disorders) | 1 (1) | 1 (1)
Cognitive Impairment (General disorders) | 1 (1) | 3 (3)
Unusual discomfort to warm temperatures (General disorders) | 1 (1) | 0 (0)
Increased Appetite (General disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight Gain (General disorders) | 1 (1) | 1 (1)
Dizziness/Lightheadedness (General disorders) | 1 (1) | 6 (6)
Dry Mouth (General disorders) | 0 (0) | 11 (11)
Consitpation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 2 (2)
Hot flashes (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No